CLINICAL TRIAL: NCT00395447
Title: Prospective Assessment of the Complication Rate After Device Replacement Due to ERI, Advisory or Upgrade
Brief Title: REPLACE: Implantable Cardiac Pulse Generator Replacement Registry
Acronym: REPLACE
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REPLACE
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Device Replacement; Elective Replacement (ERI); Device Advisory; Device Upgrade; Postoperative Complications
Keywords: Cardiac Pacemaker; Defibrillator; Replacement; Upgrade
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Straight-forward Device Replacement: Subject with a straight-forward device replacement without lead revisions or additions.
  Interventions: Procedure: Straight-forward Device Replacement
- Device Replacement with Upgrade: Subjects with a device replacement and planned lead upgrade, revision, or addition.
  Interventions: Procedure: Device Replacement with Upgrade

INTERVENTIONS:
Procedure: Straight-forward Device Replacement
  Groups: Straight-forward Device Replacement
Procedure: Device Replacement with Upgrade
  Groups: Device Replacement with Upgrade

SUMMARY:
The objective of this study is to prospectively estimate the all-cause complication rates at 6-months for patients undergoing generator replacement due to elective replacement indicator (ERI), advisory, or upgrade without a planned system modification or with a planned system modification. Secondarily, this study aims to compare the influence of baseline variables contributing to the all-cause complication rates for subjects undergoing generator replacement.

DETAILED DESCRIPTION:
Device replacements occur for many reasons, including elective replacement indication (ERI), manufacturer advisory, and upgrade.

Recently pacemaker and implantable cardioverter (ICD) advisories have created a dilemma for both physicians and patients. While the risk of device malfunction is low, replacement rates following an advisory are usually high and complication rates following device replacement are not widely known. One retrospective analysis of ICD advisories in Canada reported an 18.3% replacement rate, and subsequent 8.1% complication rate directly related to the replacement.

Device replacements also occur in order to upgrade an existing system. Clinical studies have shown that cardiac resynchronization therapy (CRT) significantly reduces all-cause mortality and hospitalization in patients with advanced heart failure (HF). As a result of expanding indications for this therapy, many standard ICD patients are being upgraded to CRT-D systems. Complication rates related to upgrades of these systems are also not widely known.

To our knowledge, the risk of complications following a device replacement has not been studied prospectively in any patient population. Limited data are available to guide physicians when weighing the risks and benefits of device replacement.

This is a prospective multi-center study. 1750 patients at 100 clinical sites will be enrolled prior to generator replacement. Patients will be implanted and followed for 6 months to assess any complications related to the replacement procedure.

Patients with any legally marketed device for explant can be enrolled. The replacement device can be from any manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Is able to give informed consent
* Is identified for generator replacement without system modification or generator replacement including planned system modification, regardless of generator manufacturer
* Is clinically stable to tolerate the surgical procedure
* Age 18 years or greater
* Is geographically stable and able to return to the investigational site for follow-up care through the six-month visit

Exclusion Criteria:

* Inability or unwillingness to give informed consent
* Current system infection requiring generator explantation or lead extraction
* Generator replacement requiring planned lead extraction
* Participating in another cardiovascular investigational drug or device registry
* A life expectancy of less than six months
* Expected to receive a heart transplant within 6 months
* All vulnerable subjects as defined by the FDA Office of Human Research Protection or the local IRB providing oversight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with device replacement procedures at study sites
Sampling Method: Probability Sample
Enrollment: 1744 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Poole, MD, Principal Investigator — University of Washington
Locations (71):
- United States (71):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mesa Cardiovascular, Mesa, Arizona
  - Stanislaus Cardiology, Modesto, California
  - Desert Cardiology, Rancho Mirage, California
  - Mercy General Hospital, Sacramento, California
  - UCSD Medical Center, San Diego, California
  - UCSF, San Francisco, California
  - Penrose Hospital, Colorado Springs, Colorado
  - Aurora Denver Cardiology, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Manatee Memorial, Bradenton, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Baptist Jacksonville, Jacksonville Beach, Florida
  - Mt. Sinai Medical Center, Miami Beach, Florida
  - Wuesthoff Hospital, Rockledge, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Florida Medical Center, Zephyrhills, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Clinic, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Central Baptist, Lexington, Kentucky
  - Louisiana Heart, Lafayette, Louisiana
  - Tulane University, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Midatlantic Cardiovascular Associates, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Shady Grove Adventist, Rockville, Maryland
  - Tufts University, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - New England Cardiovascular Specialists, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - North Shore Medical Center, Salem, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - Forrest General Hospital, Hattiesburg, Mississippi
  - Mid America Heart, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Heart Consultants Omaha, Omaha, Nebraska
  - Alegent Hospitals, Omaha, Nebraska
  - Creighton University, Omaha, Nebraska
  - St. Barnabas, West Orange, New Jersey
  - Buffalo Heart Group, Buffalo, New York
  - St. Luke's Roosevelt Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland, Cleveland, Ohio
  - Heart and Vascular Center, MetroHealth MC, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OU Medical Center Presbyterian, Oklahoma City, Oklahoma
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Sacred Heart Medical Center, Eugene, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Abington Medical Specialists, Abington, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Pee Dee Cardiology, Florence, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Amarillo Heart, Amarillo, Texas
  - Christus Spohn, Corpus Christi, Texas
  - UT Southwestern, Dallas, Texas
  - Heart Center of North Texas, Fort Worth, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - CAMC Memorial Hospital, Charleston, West Virginia

REFERENCES:
- [Derived] Chung MK, Holcomb RG, Mittal S, Steinberg JS, Gleva MJ, Mela T, Uslan DZ, Mitchell K, Poole JE; REPLACE Investigators. REPLACE DARE (Death After Replacement Evaluation) score: determinants of all-cause mortality after implantable device replacement or upgrade from the REPLACE registry. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1048-56. doi: 10.1161/CIRCEP.114.001671. Epub 2014 Sep 14. PMID 25221331
- [Derived] Uslan DZ, Gleva MJ, Warren DK, Mela T, Chung MK, Gottipaty V, Borge R, Dan D, Shinn T, Mitchell K, Holcomb RG, Poole JE. Cardiovascular implantable electronic device replacement infections and prevention: results from the REPLACE Registry. Pacing Clin Electrophysiol. 2012 Jan;35(1):81-7. doi: 10.1111/j.1540-8159.2011.03257.x. Epub 2011 Nov 11. PMID 22077194
- [Derived] Poole JE, Gleva MJ, Mela T, Chung MK, Uslan DZ, Borge R, Gottipaty V, Shinn T, Dan D, Feldman LA, Seide H, Winston SA, Gallagher JJ, Langberg JJ, Mitchell K, Holcomb R; REPLACE Registry Investigators. Complication rates associated with pacemaker or implantable cardioverter-defibrillator generator replacements and upgrade procedures: results from the REPLACE registry. Circulation. 2010 Oct 19;122(16):1553-61. doi: 10.1161/CIRCULATIONAHA.110.976076. Epub 2010 Oct 4. PMID 20921437

RESULTS

PARTICIPANT FLOW:
Groups:
- 'Straight-forward' Device Replacement: Cohort for patients undergoing a straight-forward device replacement without any planned system modification
- Replacement With Planned System Modification: Cohort for patients undergoing device replacement that includes a planned lead addition or revision. The complication rate is defined as the percentage of patients experiencing one or more major complication.
Period: Overall Study
Arm/Group | 'Straight-forward' Device Replacement | Replacement With Planned System Modification
Started | 1031 | 713
Completed | 910 | 602
Not Completed | 121 | 111
Not completed — Death | 37 | 32
Not completed — Lost to Follow-up | 52 | 43
Not completed — Withdrawal by Subject | 24 | 19
Not completed — Withdrawl - Other (not subject) | 8 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 'Straight-forward' Device Replacement | Replacement With Planned System Modification | Total
Number analyzed (Participants) | 1031 | 713 | 1744
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (14) | 70 (13) | 70 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 389 | 172 | 561
  Male | 642 | 541 | 1183
Region of Enrollment [Number; unit: participants]
  United States | 1031 | 713 | 1744

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Experiencing a Complication During Generator Replacement Without a Planned Lead Revision or Addition (Straight-forward Device Replacment) or With a Planned Lead Revision or Addition (Planned System Modification)
Description: The percentage of subjects experiencing one of the pre-defined complications is presented. The percentage of subjects experincing a complication is presented separately for subjects with a straight-forward device replacment (generator replacement procedure plan did not include a lead addition or revision) and subjects with a planned system modification (generator replacement procedure plan did include a lead addition or revision).
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | 'Straight-forward' Device Replacement | Replacement With Planned System Modification
Number analyzed (Participants) | 1031 | 713
Percentage of participants (%) | 10.8 [9.9 to 12.8] | 20.9 [18.0 to 24.1]

ADVERSE EVENTS:
Arm/Group | 'Straight-forward' Device Replacement | Replacement With Planned System Modification
Serious Adverse Events (participants affected / at risk) | 0/1031 | 0/713
Other Adverse Events (participants affected / at risk) | 0/1031 | 0/713

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained from BIOTRONIK or PharmaLink concerning the research ideas used in this study and all information obtained under or concerning this study is considered BIOTRONIK property. Investigator will maintain such information in confidence and not release it to anyone without written consent from BIOTRONIK or prior public disclosure, with the exception of information required by law or regulations to be disclosed to the reviewing IRB, the patient, or the FDA.